CLINICAL TRIAL: NCT01622426
Title: Tolerance to a New Free Amino Acid-based Formula in Children With IgE or Non-IgE-mediated Cow's Milk Allergy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RBC-100790
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Cow's Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- New formula IgE mediated testing (Active Comparator): Children with IgE-mediated CMA performed oral food challenge with the new formula
  Interventions: Dietary Supplement: tolerance to a new aminoacid based formula; Dietary Supplement: Amino acid formula
- New formula non-IgE-mediated testing (Active Comparator): Children with non-IgE-mediated CMA performed oral food challenge with the new formula
  Interventions: Dietary Supplement: tolerance to a new aminoacid based formula; Dietary Supplement: Amino acid formula

INTERVENTIONS:
Dietary Supplement: tolerance to a new aminoacid based formula — Every 20 minutes, successive doses (0.1, 0.3, 1, 3, 10, 30 and 100 mL) of placebo (the commercially available Aaf Neocate, Nutricia, Milan, Italy) or of the study formula (Sineall, Humana, Milan, Italy) were administered.
  Other Names: Sineall
Dietary Supplement: Amino acid formula — Every 20 minutes, successive doses (0.1, 0.3, 1, 3, 10, 30 and 100 mL) of placebo (the commercially available Aaf Neocate, Nutricia, Milan, Italy) or of the study formula (Sineall, Humana, Milan, Italy) were administered.
  Other Names: Sineall

SUMMARY:
The investigators aim to assess the tolerance to a new commercially available Aaf in children affected by IgE- or non-IgE-mediated CMA.

DETAILED DESCRIPTION:
Prospective controlled study including pediatric patients (≤14 years of age) with a recent diagnosis of IgE- or non-IgE-mediated CMA, confirmed by positive oral food challenge or anaphylaxis in the 2 months prior to enrollment and under good clinical control. Children with concomitant chronic systemic diseases, congenital cardiac defects, active tuberculosis, autoimmune diseases, immunodeficiency, chronic inflammatory bowel diseases, celiac disease, cystic fibrosis, metabolic diseases, lactose intolerance, malignancy, chronic pulmonary diseases, malformations of the gastrointestinal tract, gastroesophageal reflux disease non-food allergy-related, suspected eosinophilic gastrointestinal disorders, were excluded. At the first evaluation, the clinical history, information on allergic disease and baseline clinical conditions were assessed by 3 experienced pediatric allergists and the child was invited to participate in the study. At least one parent of each subject provided written informed consent. Children with atopic dermatitis were included if it was under sufficient control to allow recognition of a positive response to the challenge. Infants and children using a betablocker within 12 hours of the challenge, and short-acting, medium-acting, or long-acting antihistamines more than once within 3, 7, or 21 days of DBPCFC, respectively, or oral steroids within 21 days of oral food challenge were excluded from study. Adverse events were recorded throughout the study.

Food allergy screening tests Measurement of serum specific IgE against CMP (alpha-lactalbumin, ALA; beta-lactoglobulin, BLG; and casein); skin prick tests (SPT) with whole milk, CMP, placebo formula (another commercially available Aaf, Neocate, Nutricia, Milan, Italy) and study formula (Sineall, Humana, Milan, Italy); and atopy patch tests (APT) with whole milk, placebo and study formula, were performed on all patients.

Serum samples from patients were analysed for specific IgE antibody titers against CMP using a commercially available kit (CAP-RAST, Pharmacia Diagnostics AB, Uppsala Sweden). The detection limit of the system was 0.35 kU/L IgE. Subjects were deemed sensitised if their specific IgE levels exceeded the detection limit.

Skin prick tests were performed using a 1-mm single peak lancet (ALK, Copenhagen, Denmark), with histamine dihydrochloride (10 mg/ml) and isotonic saline solution (NaCl 0.9%) as positive and negative control, respectively. Reactions were recorded on the basis of the largest diameter (in millimetres) of the wheal and flare at 15 min. The SPT result were considered "positive" if the wheal was 3 mm or larger, without reaction of the negative control.

Atopy patch tests were performed as previously reported. Briefly, we used 1 drop (50 μl) of fresh milk put on filter paper and applied with adhesive tape to the unaffected skin of the child's back, using 12-mm aluminium cups (Finn Chambers on Scan pore; Epitest Ltd Oy, Tuusula, Finland). Isotonic saline solution was the negative control. The occlusion time was 48 h and results were read 20 min and 24 h after removal of the cups. To exclude false positive reactions, we also tested allergens in a 1:10 solution. Seventy-two hours after the start of the test, reactions were classified as follows: - negative; +/- doubtful: erythema only; + weak positive: erythema, slight infiltration, papules; ++ strong positive: erythema, infiltration, papules, little vesicles; +++ very strong positive: erythema, large confluent vesicles in bubbles. Children and their families were requested to report any delayed skin reaction that was noticed after this time. Irritant or doubtful reactions, including sharply demarcated confluent erythema, or reactions confined to margins without infiltration, were deemed negative.

Oral food challenge All food challenges were performed in a double blind placebo controlled food challenge (DBPCFC) manner, and took place in the outpatients clinic on 2 separate days with a one week interval, as previously reported. A 7-day period of strict elimination of CMP and other suspected food allergens preceded the DBPCFC. The results were assessed simultaneously by 3 experienced pediatric allergists in each center. Randomization and preparation of the challenges were performed by clinical dieticians not directly involved in the study; a separate computer-generated randomization list of participant numbers that indicated in order in which each study formula should be offered in the DBPCFC challenge was created.

Briefly, every 20 minutes, successive doses (0.1, 0.3, 1, 3, 10, 30 and 100 mL) of placebo (the commercially available Aaf Neocate, Nutricia, Milan, Italy) or of the study formula (Sineall, Humana, Milan, Italy) were administered. Full emergency equipment and drugs (epinephrine, antihistamines, and steroids) were at hand. Study subjects were scored for nine items divided into four main categories (general, skin, gastrointestinal, and respiratory) on a 0- to 3-point scale (0, none; 1, light; 2, moderate; and 3, severe). If at least two of the 3 specialists independently scored any item at level 3, or 2 (or more) items at level 2, the test result was considered positive. The patients were observed for 2 h after the final dose, and then discharged. In the case of a positive DBPCFC, at any testing dose, the patient remained under observation until after symptoms resolved. If patients did not show any symptoms within the first 24 hours, to assess long-term tolerance and reveal any false-negative results to the challenges, parents were advised to administer to the patients one single top dose of the tested formula (verum or placebo) everyday at home for seven days (7-day home feeding period). Participants' parents recorded in a daily diary volume of formula consumed; presence and severity of vomiting, diarrhea, rash, runny nose, wheezing, or any other symptoms (rated as mild, moderate, or excessive); and number of bowel movements. If any symptoms occurred during this period, the patients returned to the outpatient clinic on the same day. The investigator completed a final evaluation at the end of the 7-day home feeding period. After 7-day home feeding period of verum or placebo administration, the patients were examined and the parents interviewed at the Centers. To rule out false-negative challenge result parents were asked to contact the Center if any symptoms occurred in the following 7 days after the DBPCFC procedures. The challenge was considered negative if the patient tolerated the entire challenge, including the observation period.Markers of intestinal mucosa inflammation The fecal concentration of calprotectin (FC) and of eosinophilic cationic protein (ECP) was determined 24 hours before and 7 and 14 days after DBPCFC to evaluate the occurrence of even subclinical intestinal mucosa inflammation in response to Aaf exposure. Stool samples were collected, stored at -20°C and analyzed at the end of the study by a researcher blinded to the results of DBPCFC. Fecal calprotectin levels were measured by a highly sensitive enzyme-linked immunosorbent assay (ELISA, Calprest®, Eurospital, Italy).

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (≤14 years of age) with a recent diagnosis of IgE- or non-IgE-mediated CMA, confirmed by positive DBPCFC or anaphylaxis in the 2 months prior to enrollment and under good clinical control.

Exclusion Criteria:

* Children with concomitant chronic systemic diseases
* Congenital cardiac defects
* Active tuberculosis
* Autoimmune diseases
* Immunodeficiency
* Chronic inflammatory bowel diseases
* Celiac disease
* Cystic fibrosis
* Metabolic diseases
* Lactose intolerance
* Malignancy
* Chronic pulmonary diseases
* Malformations of the gastrointestinal tract
* Gastroesophageal reflux disease non-food allergy-related
* Suspected eosinophilic gastrointestinal disorders, were excluded.

Ages: 1 Month to 168 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2008-10; Primary Completion 2010-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Tolerance to a new free amino acid-based formula in children with IgE or non-IgE-mediated cow's milk allergy | about 2 year
  Consecutive patients affected by IgE- or non-IgE-mediated CMA, aged ≤ 14 years, were enrolled. Oral food challenge was carried out with increasing doses of the new Aaf (Sineall, Humana, Milan, Italy), using validated Aaf as placebo. Fecal concentrations of calprotectin (FC) and eosinophilic cationic protein (ECP) were monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Berni Canani, MD, PhD, Principal Investigator — Federico II University
Locations (1):
- University of Naples Federico II, Naples, Naples, Italy

REFERENCES:
- [Derived] Berni Canani R, Nocerino R, Leone L, Di Costanzo M, Terrin G, Passariello A, Cosenza L, Troncone R. Tolerance to a new free amino acid-based formula in children with IgE or non-IgE-mediated cow's milk allergy: a randomized controlled clinical trial. BMC Pediatr. 2013 Feb 18;13:24. doi: 10.1186/1471-2431-13-24. PMID 23418822